CLINICAL TRIAL: NCT03802058
Title: Concurrent Nab--paclitaxel/Carboplatin and Thoracic Radiotherapy in Inoperable Stage III Squamous Cell Lung Cancer
Brief Title: Concurrent Nab-P/Carboplatin and Thoracic Radiotherapy in Squamous Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted because enrollment was too slow
Sponsor: Wuhan University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, director of Department of Radiation and Medical Oncology, Zhongnan Hospital, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nab-P RT
Record Dates: First submitted 2019-01-06; First posted 2019-01-14 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel (Experimental): Nab-paclitaxel and carboplatin for Injection; thoracic radiation therapy
  Interventions: Drug: Nab-paclitaxel; Drug: Carboplatin; Radiation: Thoracic radiation therapy

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel 40mg/m2 for Injection weekly
  Other Names: Nab-P
Drug: Carboplatin — Carboplatin AUC=2 for Injection weekly
  Other Names: CBP
Radiation: Thoracic radiation therapy — Thoracic radiation therapy 60-66Gy/30-33 fractions,both three-dimensional conformal and intensity modulated radiation therapy are allowed
  Other Names: RT

SUMMARY:
Nab-paclitaxel and carboplatin showed better treatment response compared with cremophor-based paclitaxel and carboplatin as first-line therapy in advanced non-small cell lung cancer, especially for squamous cell cancer. This study is conducted to evaluate the efficacy and safety of nab-paclitaxel, carboplatin and concurrent radiotherapy in patients with local advanced inoperable squamous cell lung cancer.

DETAILED DESCRIPTION:
This study was conducted to explore the efficacy and safety of concurrent concurrent nab-paclitaxel, carboplatin and thoracic radiotherapy in inoperable local advanced squamous cell lung cancer. Patients will be given nab-paclitaxel weekly at a dose of 40mg/m2, in combination with carboplatin (AUC 2) weekly during concurrent chemoradiotherapy. Thoracic radiation was administered at a dose of 60-66 Gy/30-33 fractions, both 3 dimensional conformal and intensity modulated radiation therapy are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 Years to 70 Years
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Previously untreated, histological documented, inoperable stage III squamous cell carcinoma of lung, excluding those with pericardial, pleural effusion, and those with contralateral hilar or contralateral supraclavicular lymph nodes.
* Patients must have measurable disease according to RECIST criteria, and all detectable tumor can be encompassed by radiation therapy fields.
* Patient must have adequate blood, liver, lungs and kidney function within the requirements of this study.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.
* Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Complete tumor resection, recurrent disease, or those patients eligible for definitive surgery.
* Previous chemotherapy or previous biologic response modifiers for current lung cancer.
* Patient has previously had thoracic radiation therapy.
* Prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for five years or more.
* Serious concomitant disorders that would compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
PFS (progression-free survival ) | 5 years from patient enrollment
  PFS is defined as time from the start of treatment to death, progression of disease, or the last follow-up data, whichever comes first. Progression is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. PFS will be analyzed using the Kaplan-Meier method.

SECONDARY OUTCOMES:
ORR (Overall Response Rate ) | one month after the end of all treatment
  The number of participants that achieve either a complete response (CR) or a partial response (PR). Response is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
LCR (Local Control Rate) | one month after the end of all treatment
  The number of participants that achieve either a complete response (CR) , a partial response (PR) or stable disease(SD).
OS (Overall survival) | 5 years from patient enrollment
  Overall survival is defined as time from the start of treatment until death. Overall survival will be analyzed using the Kaplan-Meier method.
Number of participants with adverse events as assessed by CTCAE v4.0 | 5 years from patient enrollment
  The adverse events(AE) is evaluated by National Cancer Institute- Common Terminology Criteria for Adverse Events(NCI -CTCAE) 4.02.
Patient quality of life (QOL) | 5 years from patient enrollment
  Measured by the Functional Assessment of Cancer Therapy - Lung (FACT-L).The total range of scores:0-144,and higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Conghua Xie, Dr, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD can be shared by all researchers who participate in this study by e-mail contact
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years after the end of the study
Access Criteria: Researchers who participate in this study